CLINICAL TRIAL: NCT04390737
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Activity of HH2853 in Patients With Relapsed/Refractory Non-Hodgkin's Lymphomas or Advanced Solid Tumors
Brief Title: Evaluate the Safety and Clinical Activity of HH2853
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH2853-G101
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: FL Lymphoma; Epithelioid Sarcoma; Peripheral T Cell Lymphoma; Advanced Solid Tumor
Keywords: Phase I/II; HH2853; PRC2; EZH 1/2 inhibitor
MeSH Terms: conditions — Lymphoma, Follicular; Sarcoma; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HH2853 administered on a BID schedule in continuous 28-day treatment cycles (Experimental): HH2853 is supplied as tables with dosage strength of 25mg and 200mg. HH2853 Tablet will be administered orally on a continuous twice daily (BID) schedule, on a flat scale of mg and not individually adjusted by weight or body surface area. A treatment cycle is defined as 28 days for the purposes of scheduling procedures and evaluations.
  All patients will be treated with HH2853 orally on a continuous BID schedule, beginning on Cycle 1 Day 1. But patients in accelerated titration (ATD) part should be administered a single dose on the first day in order to evaluate the PK of a single dose administration. Dosing is twice daily from the second day thereafter.
  Interventions: Drug: HH2853 Tablets

INTERVENTIONS:
Drug: HH2853 Tablets — Proposed daily dose (BID): 50mg, 100mg, 200mg, 400mg, 600mg, 800mg, 1000mg. It is possible for additional and/or intermediate dose levels to be added during the course of the study. Cohorts may be added at any dose level below the MTD in order to better understand safety, PK or PD.

SUMMARY:
This is an open-label, multicenter, first-in-human phase I/II study which is composed of 3 parts: phase I dose escalation, phase I dose extension and phase II. HH2853 will be administered orally on a continuous BID schedule on a continuous 28-day treatment cycle.

DETAILED DESCRIPTION:
Phase I:

Phase I dose escalation The accelerated titration (ATD) incorporated with Bayesian Optimal Interval design (BOIN) will be used to assess the DLT, safety, tolerability, MTD and furthermore, to establish the RP2D. DLT assessment is only applicable to phase I dose escalation.

Eligible patients will be enrolled in the ascending dose until MTD/RP2D is established.

Phase I dose extension During the dose escalation phase, a dose extension with additional patients will be included in order to further evaluate the tolerability, pharmacokinetics, and efficacy at doses that have been evaluated as safe. The number of patients to be enrolled in each dose extension cohort is up to 15, but the final number of dose level can be determined and the final patient number at each dose level can be adjusted slightly based on available safety, efficacy, PK, and PD data upon agreement from sponsor and investigators (e.g. safety evaluation meeting). For phase I dose extension, approximately 30 patients will be enrolled based on initial estimate, but the final total number of patients will depend on the number of dose levels extended and patient number at each dose level.

The total number of patients is estimated to be approximately 60 patients for phase I dose escalation and dose extension, but the final total number of patients will depend upon the number of dose cohorts to reach MTD/RP2D, and patient number at each dose level.

Phase II（China Only）:

Phase II is planned after the completion of phase I. Up to approximately 193 patients will be enrolled as outlined below:

* Cohort 1: Relapsed/Refractory FL (n≈56)
* Cohort 2: Epithelioid sarcoma (n≈77)
* Cohort 3: Relapsed/Refractory PTCL, other relapsed/refractory Non-Hodgkin's lymphomas with EZH2 mutation, or advanced solid tumors with specific genetic alterations, including EZH2 mutation, INI1 deficiency, BAP1 deficiency, ARID1A mutation, or/and SMARCA4 mutation (n≈60)

ELIGIBILITY:
Inclusion criteria:

1. Provided signed written informed consent prior to initiation of any study-related procedures;
2. Males and females ≥ 18years of age at the time of consent are obtained (or meet the country's regulatory defined adult legal age);
3. Tumor type criteria:

The specific requirements for specific subtypes of recurrent/refractory non Hodgkin's lymphoma (NHL) confirmed by histology are as follows:

Histologically confirmed follicular lymphoma (FL) that has been treated with at least two lines of systemic therapy (at least one regimen based on anti-CD20 monoclonal antibodies) according to GELF criteria or as determined by researchers (Grade 1-3a); Relapsed/refractory diffuse large B-cell lymphoma - non-specific (DLBCL NOS, 2016 World Health Organization Lymphoma Classification) that has received at least two treatment regimens in the past (at least one with CD20 monoclonal antibody as the main treatment, with a maximum number of treatment lines<5), and is not a candidate for salvage treatment or autologous/allogeneic stem cell transplantation.

Relapsed/refractory clinicopathologically documented PTCL with at least 1 line of prior systemic treatment (maximum <5 lines). Solid tumors that meet the following criteria:

1. Histologically or cytologically documented advanced recurrent or metastatic solid tumor.
2. Phase I dose escalation: Measurable or evaluable lesions by RECIST v1.1 in at least 1 site; phase I dose extension and phase II: Measurable target lesions by RECIST v1.1 in at least 1 site. (Lesions that have been treated with radiotherapy or other local treatment are generally considered unmeasurable unless there is definite progression of the lesion.)
3. Patients must have disease not amenable to surgery, radiation, or combined modality therapy with curative intent. One of the following criteria should be met.

Patients must experience at least one prior standard therapy. Disease progression occurred on or after last line of therapy, or intolerant to last line of therapy (maximum ≤3 lines, Patients without treatment options available known to provide clinical benefit are also eligible upon agreement from investigator and sponsor) There is no approved therapy, or for which standard therapy is unsuitable or refused by patients after being fully informed.

For epithelioid sarcoma in Phase I and Phase II cohort 2:

1. Confirmed by local histology or cytology
2. Patients with unresectable locally delayed or metastatic epithelioid sarcoma who have undergone treatment (including those who have failed treatment and developed intolerable toxicity).

For solid tumors in Phase I and Phase II queue 3:

1. Confirmed by local pathology as advanced recurrent or metastatic solid tumor.
2. Patients must have disease not amenable to surgery, radiation, or combined modality therapy with curative intent 4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1; 5. Availability of archival tissue within three years 6. Relapsed/Refractory FL, Epithelioid sarcoma, relapsed/refractory PTCL, other relapsed/refractory non-Hodgkin's lymphomas with EZH2 mutation, and advanced solid tumors with specific genetic alterations, including EZH2 mutation, INI1 deficiency, BAP1 deficiency, ARID1A mutation, or/and SMARCA4 mutation 7. Predicted life expectancy of ≥ 3 months; 8. Patient must meet the following laboratory values: 1.Serum total Bilirubin ≤ 1.5 x ULN or ≤ 3.0 mg/dL for patients with Gilbert's syndrome 2.AST/SGOT and ALT/SGPT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present 3.24-hour creatinine clearance (calculated* or measured value**)≥ 50 mL/min 4.Platelets ≥ 1 x LLN (no Platelet transfusion for 7 days prior to screening) 5.Hemoglobin (Hgb) ≥ 9 g/dL 6.Absolute Neutrophil Count (ANC) ≥ 1.0 x 10^9/L 7.Adequate coagulation function: International normalized ratio (INR) <1.3 (or <3.0 on anticoagulants) 9. Measurable lesion

Exclusion Criteria:

1. Any cancer-directed therapy within 28 days or five half-lives prior to first dose; Small molecule anticancer therapy within 2 weeks or five half-lives; Local radiotherapy within 14 days of first dose.
2. Symptomatic CNS metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.
3. Patients with prior transplant are excluded;
4. Major surgery within 4 weeks prior to first dose;
5. A prohibited medication or expected to require any of these medications during treatment with study drug within 2 weeks of first dose;
6. HIV (human immunodeficiency virus) infection, active hepatitis B or hepatitis C patients (HBsAg positive patients with HBV (hepatitis B virus) DNA ≥ 10^3 copies or ≥ 200 IU/mL; HCV antibody test results are positive, and HCV (hepatitis C virus) RNA PCR test results are positive).
7. Concomitant malignancies or previous malignancies
8. Concurrent use of therapeutic warfarin is allowed. However, anticoagulants that do not have reversal agents available are prohibited except low molecular weight heparin and direct oral anticoagulants.
9. Any toxicities from prior treatment that have not recovered to ≤ CTCAE Grade 1
10. There were ≥ 3 lesions with punctate bleeding, any active bleeding, intratumoral bleeding, known bleeding tendencies, or treatment with antiplatelet/antithrombotic drugs.
11. Gastrointestinal condition which could impair absorption of study medication;
12. Psychological, familial, sociological or geographical conditions that do not permit compliance with the protocol;
13. Cardiac exclusion criteria:

1.History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 3 months prior to first dose of study drug; 2.Fridericia's corrected QT interval (QTcF) > 450 ms (for male) and > 470 ms (for female) on ECG conducted during screening; 3.Congenital long QT syndrome, or any known history of torsade de pointes (TdP), or family history of unexplained sudden death; 4.History or current evidence of serious uncontrolled ventricular arrhythmias; 5.Symptomatic congestive heart failure (Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system) within the previous 3 months; 6.Left ventricular ejection fraction (LVEF) < 50%; 14. Any evidence of serious active infections requiring antibiotics; 15. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug or their excipients; 16. Pregnant or breast-feeding female; 17. Contraception: 18. Other serious illness or medical conditions at the Investigator's discretion, that may influence study results 19. Previously received treatment with EZH2 or EZH1/2 inhibitors. 20. Grade 3b FL or evidence of transformation to invasive lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated Dose (MTD) | 28-day treatment cycles
  Determine MTD of HH2853
Recommended phase II dose (RP2D) | 28-day treatment cycles
  Determine RP2D of HH2853
Adverse events assessed according to NCI-CTCAE V5.0 | 28-day treatment cycles
  Evaluate the safety of HH2853
Dose limiting toxicities (DLT) | 28-day treatment cycles
  Evaluate the tolerability of HH2853
Objective response rate (ORR） | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853

SECONDARY OUTCOMES:
AUClast | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
AUCinf | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
Cmax | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
Tmax | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
CL/F | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
Vz/F | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
Terminal half-life (T1/2) | 28-day treatment cycles
  Characterize the pharmacokinetic profile of HH2853
Duration of response (DoR) | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853
Progression-free survival (PFS) | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853
Disease control rate (DCR) | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853
Time to response (TTR) | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853
Time to progression (TTP) | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853
Clinical Outcome | 28-day treatment cycles
  Explore the association between potential biomarker and the clinical outcome

OTHER OUTCOMES:
Overall survival (ORR） | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853
Change in tri-methylation of Histone H3K27 (H3K27me3) | 14-day treatment
  Assss the pharmacodynamic response
Biomarker Status | 28-day treatment cycles
  Explore the relationship between the alteration status of biomarker and treatment efficacy
Overall survival (OS) | 28-day treatment cycles
  Assess the preliminary efficacy of HH2853

CONTACTS AND LOCATIONS:
Overall Officials: Fugen Li, Study Director — Haihe Biopharma Co., Ltd.
Locations (24):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - NEXT Oncology, San Antonio, Texas
- China (20):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangdong
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Liaoning Cancer Hospital&Institute, Shenyang, Liaoning
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - Linyi Tumor Hospital, Linyi, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Sun Yat-Sen University Cancer Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in China, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.haihepharma.com/
Supporting Information: Study Protocol
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in China
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://www.icmje.org/

REFERENCES:
- [Derived] Fan Z, Wang J, Liu D, Shen L, Fang M, Johnson P, Tun H, Sommerhalder D, Yang J, Yang Y, Munozi J, Zhu J, Gao T, Li Z, Li X, Ma Q, Lv C, Yu S, Li F, Song Y, Gong J. Safety and efficacy of HH2853, a novel EZH1/2 dual inhibitor, in patients with refractory solid tumours or non-Hodgkin lymphomas: a phase I study. EClinicalMedicine. 2025 Aug 7;86:103398. doi: 10.1016/j.eclinm.2025.103398. eCollection 2025 Aug. PMID 40821900
- [Derived] Hong H, Chen Z, Zhang M, Peng Z, Shen J, Shuang Y, Zhou H, Guo H, Huang H, Li F, Qian Z, Liu L, Wang L, Yang W, Zhang L, He P, Qian S, Li F, Li M, Lin T. A multicenter, open-label, single-arm, phase Ib clinical trial of HH2853 treatment in patients with relapsed and/or refractory peripheral T-cell lymphoma. J Hematol Oncol. 2025 Apr 27;18(1):50. doi: 10.1186/s13045-025-01697-z. PMID 40289142